CLINICAL TRIAL: NCT01544907
Title: Prospective Randomized Trial Comparing Drug Eluting Balloon Angioplasty Versus Conventional Percutaneous Transluminal Angioplasty Balloon for the Treatment of Hemodialysis Arterio-Venous Fistula or Arterio-Venous Graft Stenoses
Brief Title: Prospective Randomized Trial Comparing DEB Versus Conventional PTA for the Treatment of Hemodialysis AVF or AVG Stenoses
Acronym: DEBAPTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Singapore General Hospital (Other)
Collaborators: National Medical Research Council (NMRC), Singapore (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEBAPTA
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-11

CONDITIONS: Stenosis of Arteriovenous Dialysis Fistula; Arteriovenous Graft Stenosis
Keywords: Drug Eluting Balloon; Arteriovenous fistula or graft stenosis
MeSH Terms: conditions — Arteriovenous Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Conventional PTA only (Active Comparator): Treatment Arm 1- Conventional PTA only
  The conventional balloon is used and the diameter of the balloon should be the same or oversized by 1mm the diameter of the reference vessel.
  An inflation device with a pressure gauge is used to inflate up to manufacturers' stated burst pressure. The duration of balloon inflation will be 2 minutes.
  At the end of the first angioplasty, an AVFistulogram/AVGraftogram will be obtained to document results. If there is residual stenosis of >30%, a repeat angioplasty using the same balloon or another appropriately oversized balloon by 1mm will be used for an additional 2 minutes. A final angiogram will be obtained for documentation.
  Interventions: Device: Conventional PTA
- Drug Eluting Balloon (DEB) (Experimental): Treatment arm 2 - Conventional Balloon with DEB
  A Conventional balloon is used to pre-dilate the target lesion. The DEB of a similar diameter to the conventional balloon used is then inflated across the stenosis. An inflation device with a pressure gauge is used to inflate up to manufacturers' stated burst pressure. The duration of balloon inflation will be 1 minute. A final angiogram will be obtained for documentation. The drug coated on the DEB is Paclitaxel.
  Interventions: Device: Drug Eluting Balloon (DEB)

INTERVENTIONS:
Device: Conventional PTA — Use of conventional balloon for angioplasty only
  Other Names: REEF angioplasty balloon (Manufacturer Medtronic)
  Arms: Conventional PTA only
Device: Drug Eluting Balloon (DEB) — Use of DEB after conventional balloon angioplasty
  Other Names: IN.PACT ADMIRAL Paclitaxel-eluting Balloon (Medtronic)
  Arms: Drug Eluting Balloon (DEB)

SUMMARY:
A prospective randomized trial comparing the efficacy of drug eluting balloon angioplasty versus conventional percutaneous transluminal angioplasty balloon for the treatment of hemodialysis arterio-venous fistula or arterio-venous graft stenoses in reducing late luminal loss and restenosis rates, while prolonging primary and secondary patencies.

DETAILED DESCRIPTION:
Introduction:

Neointimal hyperplasia is the main cause of hemodialysis access [arterio-venous fistula (AVF) or graft (AVG)] dysfunction and thrombosis. Although endovascular techniques like percutaneous transluminal angioplasty (PTA), catheter directed thrombolysis, mechanical thrombectomy or bare metal stenting, may salvage the access, long term patency remains dismal due to recurrent stenosis from neointimal hyperplasia.

Drug Eluting Balloon (DEB) is effective in inhibiting neointimal hyperplasia for treatment of coronary in-stent restenosis since 2006 and more recently in femoropopliteal arteries, reducing restenosis rates and prolonging patency.

Specific Aim:

To determine the efficacy of DEB in reducing restenosis rates and prolonging the patency of AVFs/AVGs compared to PTA.

Hypothesis:

DEB is superior to PTA in reducing late luminal loss and restenosis rates, while prolonging primary and secondary patencies.

Methodology:

Prospective, randomized clinical trial with study population comprising of patients with dysfunctional AVFs/AVGs due to underlying stenoses. The patients will be randomized to receive either DEB or PTA.

The 6-month late luminal loss will be primary endpoint. The secondary endpoints of restenosis rate, primary and secondary patencies, will also be determined.

Major Clinical Significance:

Hemodialysis access failures constitute significant morbidity and costs to patient and healthcare system. Maintaining access patency consumes significant resources and constitutes a significant portion of the work of vascular surgeons, nephrologists and interventional radiologists.

Any strategy that reduces access failure or prolonging access lifespan will be beneficial. If DEB is proven to be superior to PTA, there will be a paradigm shift in management of hemodialysis access failures from restenosis - similar to how DEB has changed practice in managing coronary artery in-stent restenosis.

ELIGIBILITY:
Inclusion Criteria:

1. Upper limb or groin AVF/AVG
2. The AVF/AVG is > 3 months old.
3. Native vessel measures between 4 to 7 mm diameter (corresponding to the sizes of available DEBs).
4. The fistula or graft must not be thrombosed.
5. Able to cross with guide wire
6. Platelet count >50,000/l (platelet infusion if <100,000/l)
7. PT/PTT not more than 3 seconds above normal (FFP infusion for abnormal PT/PTT)

Exclusion Criteria:

1. Uncorrectable coagulopathy (despite transfusion) or hypercoagulable state.
2. Evidence of systemic infection or a local infection associated with the fistula or graft.
3. The patient is < 21 years of age.
4. The patient is pregnant.
5. Patient is enrolled in another investigational study
6. Patient has comorbid conditions that may limit their ability to comply with the follow-up requirement.
7. Life expectancy < 6 months

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2012-01; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Late luminal loss | 6 months
  Late luminal loss is defined as the difference between the minimum lumen diameters after angioplasty and at the end of the 6-month follow-up angiogram.

SECONDARY OUTCOMES:
Restenosis rate | 6 months
  Restenosis rate is defined as the incidence of stenosis ≥50% of the diameter of the reference vessel segment.
Primary patency | 6 months
  Primary patency is defined as the interval from balloon angioplasty until the next access thrombosis or repeated intervention to maintain access function, or until access abandonment if no interval intervention. It ends with treatment of a lesion anywhere within the access circuit, from the arterial inflow to the superior vena cava-right atrial junction.
Primary assisted patency | 6 months
  Primary assisted patency is defined as the interval from balloon angioplasty until access thrombosis or a surgical intervention that excludes the treated lesion from the access circuit. Examples include percutaneous treatments of either restenosis/occlusion of the previously treated lesion or a new arterial or venous outflow stenosis/occlusion (excluding access thrombosis). It ends with percutaneous thrombolysis/thrombectomy or simple surgical thrombectomy.
Secondary patency | 6 months
  Secondary patency is defined as the interval after balloon angioplasty until the access is surgically declotted, revised or abandoned because of inability to treat the original lesion, choice of surgeon, transplant, loss to follow-up, etc. Examples include thrombolysis and percutaneous thrombectomy, as well as multiple repetitive treatments.
Anatomic success | Immediate post procedure
  Anatomic success is defined as <30% residual stenosis diameter measured immediately after angioplasty.
Clinical success | Immediate post procedure
  Clinical success is defined as an improvement from baseline in the clinical or hemodynamic parameter (e.g., blood flow, venous pressures) that was the initial indicator of fistula/ graft dysfunction.
Procedural success | Immediate post procedure
  Procedural success is defined as the combination of anatomic success and clinical success.

CONTACTS AND LOCATIONS:
Overall Officials: Farah G Irani, MBBS,FRCR, Principal Investigator — Singapore General Hospital
Locations (1):
- Singapore General Hospital, Singapore, Singapore